CLINICAL TRIAL: NCT02706769
Title: A Double-blind Randomised Parallel Group Trial of Paracetamol Versus Placebo in Conjunction With Strong Opioids for Cancer Related Pain
Brief Title: Paracetamol Versus Placebo in Conjunction With Strong Opioids for Cancer Pain
Acronym: PaSO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated early due to slow recruitment.
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AC15006
Record Dates: First submitted 2016-01-25; First posted 2016-03-11 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Participants will take blinded Paracetamol (as they were taking before entering the study)
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Participants will take blinded Paracetamol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Study medication contains blinded placebo
  Arms: Placebo
Drug: Paracetamol — Study medication contains blinded paracetamol
  Arms: Paracetamol

SUMMARY:
National guidelines advocate the use of paracetamol in conjunction with strong opioids for cancer pain, despite a lack of evidence for its efficacy. Work is needed to examine the analgesic benefit of paracetamol in this large patient group. The investigators aim to establish if paracetamol in combination with strong opioids provides superior analgesia for cancer related pain over strong opioids alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years and over
2. Under palliative care/oncology service review
3. Diagnosis of incurable cancer
4. Clinician-predicted life expectancy >2 months
5. Anticipated to be clinically stable for duration of study involvement
6. Receiving daily regular strong opioids
7. Able to take study drug/placebo in its current form
8. Prescribed and taking paracetamol 1g four times a day
9. Average pain >3 and <9 in past 24 hours
10. Able to provide written informed consent
11. Able to complete necessary assessments required as part of the trial
12. Average NRS pain score stable (ie. maximum range of 1 point) for the three consecutive days prior to randomisation

Exclusion Criteria:

1. Pain which the clinician deems to be unstable
2. Clinically significant renal or liver disease
3. Weight less than 50kg
4. Those whose pain is expected to change during the course of the study as a result of oncological or other treatments
5. Co-enrolment in other drug trials
6. Known to be pregnant or breast-feeding at the time of recruitment
7. Previously enrolled in this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a 30% increase in total Brief Pain Inventory between day 0 and day 14 in the active drug group versus the placebo group. | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided